CLINICAL TRIAL: NCT03156608
Title: Evaluation of the Novii External Fetal Monitoring Device: A Prospective, Randomized Comparison
Brief Title: Novii External Fetal Monitoring Device
Acronym: Novii
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Michael Sean Esplin, Professor, Division of Maternal Fetal Medicine, Intermountain Health Care, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1050411
Record Dates: First submitted 2017-03-14; First posted 2017-05-17 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Pregnancy Related; Fetal Distress
Keywords: External Fetal Heart Rate Monitor; Fetal Heart Rate Monitor
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Intervention Model Description: Women will be randomized to either standard monitoring with external Doppler and tocodynamometer or monitoring with the Novii Fetal ECG/EMG system using a computer generated randomization scheme through REDCap. Randomization will occur in blocks based on the subject's BMI. Women with a BMI < 30 will be randomized separate from women with a BMI > 30.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Novii Device ECG/EMG System (Experimental): These patients will have the Novii ECG/EMG system placed throughout labor and delivery, unless a provider or investigator determines that a different device (internal or external) is necessary for a better signal.
  Interventions: Device: Novii ECG/EKG System
- Standard of Care External Monitor (Active Comparator): A standard external monitor will be placed throughout labor and delivery, unless a provider or investigator determines that an internal device is necessary for a better signal.
  Interventions: Device: External fetal heart rate monitoring

INTERVENTIONS:
Device: Novii ECG/EKG System — External fetal heart rate monitoring
  Arms: Novii Device ECG/EMG System
Device: External fetal heart rate monitoring — External fetal heart rate monitoring
  Arms: Standard of Care External Monitor

SUMMARY:
This study will be conducted on women in labor. Fetal heart rate monitoring will be conducting using the Novii Fetal ECG/EMG system and comparing it to current standard of care external fetal heart rate and tocometry. These approaches will be compared with the respect to need for additional monitoring, amount of nursing intervention, cost and satisfaction of patients and healthcare providers.

DETAILED DESCRIPTION:
Interpretation of fetal heart rate monitoring during labor is one of the most common procedures performed in the practice of obstetrics. Continuous monitoring of the fetal heart rate is used to identify infants at risk for hypoxic ischemic encephalopathy and allow for intervention to prevent this terrible complication. The quality of the fetal heart rate signal is critical for appropriate interpretation of the characteristics that identify risk.

This is a prospective, randomized pragmatic trial comparing the Novii Fetal ECG/EMG system to external fetal heart rate and tocometry (standard of care) for the amount of time of interpretable fetal heart rate during labor. Randomization will occur in blocks based on BMI to control for the potential effect of BMI.

Fetal heart rate tracings from both groups of women will be reviewed in a blinded fashion by experienced Maternal Fetal Medicine (MFM) physicians who will assess the tracing for quality and interpretability. In addition, both approaches will be compared with respect to the need for additional monitoring modalities, amount of nursing intervention, cost and satisfaction of the patients and healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ≥ 18 years of age; gestational age ≥ 37 weeks
* Singleton pregnancy.
* These women will be those presenting to Labor and Delivery for one of the following:

  * Rule out labor
  * Spontaneous labor
  * Induction of labor

Exclusion Criteria:

* Age < 18 years old; multiple gestation pregnancy; gestational age < 37 weeks
* Fetal distress or vaginal bleeding prior to monitor placement
* Previous cesarean section
* Planned cesarean delivery.
* Women who are enrolled in the study but have less than 1 hour of fetal heart rate monitoring after randomization will be excluded from analysis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 218 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Amount of time in minutes with the interpretable fetal heart rate tracing during the course of labor. | Time of randomization until time of delivery (up to 48 hours)
  Quality of the fetal heart rate for each minute of tracing will be assessed visually by 2 or more blinded reviewers. For the purpose of this study, uninterpretable fetal heart rate will be defined as continuous fetal heart rate data with one or more of the following:
  1. Data is missing for more than 75% of the minute of tracing
  2. Artifact is present for more than 25% of the minute of tracing
  3. Missing data or artifact prevents determination of baseline rate
     1. > 15 seconds of continuous missing tracing
     2. Missing data is not continuous but is sufficiently frequent that the one minute segment of tracing could not be used to determine baseline rate
  The total number of interpretable minutes of fetal heart tracing and the percentage of time with interpretable fetal heart tracing over the course of labor (Number of minutes with interpretable FHR/Total number of minutes in labor) will be calculated for each patient.

SECONDARY OUTCOMES:
Quality and interpretability of the FHT in ten minute segments | Time of randomization until time of delivery (up to 48 hours)
  a. Each 10 minute segment will be deemed to be interpretable if it meets all of the following criteria: i. Sufficient data are available to determine a baseline ii. Sufficient data are available to determine the variability of the tracing iii. Sufficient data are available to identify periodic changes in the tracing (e.g. accelerations, decelerations, etc) b. For each 10 minute segment that is called Uninterpretable, the reviewer will indicate the reason for this designation by selecting one of the following options: i. Poor signal quality due to missing data ii. Poor signal quality due to artifact iii. Adequate signal quality but intrinsic fetal heart rate makes interpretation impossible (e.g. marked variability, etc.)
Number and quality of uterine contractions in each 10 minute segment: | Time of randomization until time of delivery (up to 48 hours)
  The number of uterine contractions per segment will be recorded b. Signal quality (amount of missing data or artifact) will be recorded
Number and quality of uterine contractions in each 10 minute segment: | Time of randomization until time of delivery (up to 48 hours)
  Signal quality (amount of missing data or artifact) will be recorded
Number of times fetal heart rate monitor requires adjusting: | Time of randomization until time of delivery (up to 48 hours)
  Measured by recording the number of times the nurse must adjust the monitoring system to obtain interpretable tracing
Number of times fetal heart rate monitor requires adjusting: | Time of randomization until time of delivery (up to 48 hours)
  Number of times that hand holding of the monitor is required
Need for additional monitoring devices such as change from Novii to standard monitoring devices or the use of intrauterine pressure catheter or fetal scalp electrode: | Time of randomization until time of delivery (up to 48 hours)
  Need for additional monitoring devices will be determined by the clinical care team including attending physician and/or nurses based on clinical judgment
Need for additional monitoring devices such as change from Novii to standard monitoring devices or the use of intrauterine pressure catheter or fetal scalp electrode will be recorded by clinical care team: | Time of randomization until time of delivery (up to 48 hours)
  Reason 1: Poor signal quality - missing data Reason 2: Poor signal - artifact Reason 3: Need additional information (e.g. intrauterine pressure, etc.) Reason 4: Patient preference Reason 5: Provider preference
Need for additional monitoring devices such as change from Novii to standard monitoring devices or the use of intrauterine pressure catheter or fetal scalp electrode will be recorded by clinical care team: | Time of randomization until time of delivery (up to 48 hours)
  Reason 2: Poor signal - artifact Reason 3: Need additional information (e.g. intrauterine pressure, etc.) Reason 4: Patient preference Reason 5: Provider preference
Need for additional monitoring devices such as change from Novii to standard monitoring devices or the use of intrauterine pressure catheter or fetal scalp electrode will be recorded by clinical care team: | Time of randomization until time of delivery (up to 48 hours)
  Reason 3: Need additional information (e.g. intrauterine pressure, etc.) Reason 4: Patient preference Reason 5: Provider preference
Need for additional monitoring devices such as change from Novii to standard monitoring devices or the use of intrauterine pressure catheter or fetal scalp electrode will be recorded by clinical care team: | Time of randomization until time of delivery (up to 48 hours)
  Reason 4: Patient preference Reason 5: Provider preference
Need for additional monitoring devices such as change from Novii to standard monitoring devices or the use of intrauterine pressure catheter or fetal scalp electrode will be recorded by clinical care team: | Time of randomization until time of delivery (up to 48 hours)
  Reason 5: Provider preference
Nursing time required for care: | Time of randomization until time of delivery (up to 48 hours)
  We will record the amount of time that the nurses spend at the bedside to adjust the monitor b. Nurses will record the time and reasons that they enter the room
Nursing time required for care: | Time of randomization until time of delivery (up to 48 hours)
  Nurses will record the time and reasons that they enter the room
Overall cost of care: | Hospitalization for labor, delivery, and recovery - 2-4 days
  Total charge for care from admission to Labor and Delivery to transfer to postpartum care will be recorded for all patients
Overall cost of care: | Hospitalization for labor, delivery, and recovery - 2-4 days
  Delivery type and indication
Maternal outcomes - Length of labor | Hospitalization for labor, delivery, and recovery - 2-4 days
  Length of labor recorded
Maternal outcomes - Delivery type | Hospitalization for labor, delivery, and recovery - 2-4 days
  Type of delivery recorded (e.g., vaginal, cesarean section, etc.)
Maternal outcomes - Indication for forceps/vacuum extraction or cesarean section, if performed | Hospitalization for labor, delivery, and recovery - 2-4 days
  Clinical indication for forceps/vacuum extraction or cesarean section delivery
Maternal outcomes - Estimated blood loss | Hospitalization for labor, delivery, and recovery - 2-4 days
  Amount of blood loss (cc) recorded
Maternal outcomes - Presence and severity of perineal lacerations | Hospitalization for labor, delivery, and recovery - 2-4 days
  Lacerations and degree of laceration recorded
Maternal outcomes - Intra-amniotic infection (clinical chorioamnionitis or triple I) | Hospitalization for labor, delivery, and recovery - 2-4 days
  Infections documented
Maternal outcomes - Presence of clinical endometritis | Hospitalization for labor, delivery, and recovery - 2-4 days
  Endometritis diagnosis recorded
Neonatal outcomes - APGAR Scores | Hospitalization after delivery - 2-4 days
  APGAR scores recorded at 1 minute, 5 minutes, and 10 minutes
Neonatal outcomes - Need for ICU Admission | Hospitalization after delivery - 2-4 days
  Recorded NICU admission
Neonatal outcomes - Birthweight | Hospitalization after delivery - 2-4 days
  Infant birthweight (grams)
Neonatal outcomes - Neonatal Sex | Hospitalization after delivery - 2-4 days
  Neonatal sex recorded
Patient and provider satisfaction - Patient Survey | Up to 7 days after delivery
  Satisfaction survey completed by patient after delivery of infant
Patient and provider satisfaction - Nurse Survey | Up to 7 days after delivery
  Satisfaction survey completed by nurse attending labor/delivery after delivery of infant
Patient and provider satisfaction - Attending Physician/Midwife Survey | Up to 7 days after delivery
  Satisfaction survey completed by physician/midwife attending labor/delivery after delivery of infant

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Esplin, MD, Principal Investigator — Staff Physician
Locations (4):
- United States (4):
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley Hospital, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bakker PC, Colenbrander GJ, Verstraeten AA, Van Geijn HP. The quality of intrapartum fetal heart rate monitoring. Eur J Obstet Gynecol Reprod Biol. 2004 Sep 10;116(1):22-7. doi: 10.1016/j.ejogrb.2004.01.001. PMID 15294362
- [Background] Cohen WR, Ommani S, Hassan S, Mirza FG, Solomon M, Brown R, Schifrin BS, Himsworth JM, Hayes-Gill BR. Accuracy and reliability of fetal heart rate monitoring using maternal abdominal surface electrodes. Acta Obstet Gynecol Scand. 2012 Nov;91(11):1306-13. doi: 10.1111/j.1600-0412.2012.01533.x. Epub 2012 Oct 19. PMID 22924738
- [Background] Cohen WR, Hayes-Gill B. Influence of maternal body mass index on accuracy and reliability of external fetal monitoring techniques. Acta Obstet Gynecol Scand. 2014 Jun;93(6):590-5. doi: 10.1111/aogs.12387. Epub 2014 Apr 30. PMID 24684703
- [Background] Dawes GS, Visser GH, Goodman JD, Redman CW. Numerical analysis of the human fetal heart rate: the quality of ultrasound records. Am J Obstet Gynecol. 1981 Sep 1;141(1):43-52. doi: 10.1016/0002-9378(81)90673-6. PMID 7270621
- [Background] Rooth G, Huch A, Huch R (1987) FIGO news: guidelines for the use of fetal monitoring. Int J Gynaecol Obstet 25:159-167